CLINICAL TRIAL: NCT03100006
Title: A Phase Ib/IIa Clinical Trial to Evaluate the Safety and Activity of Oregovomab and Nivolumab as a Combinatorial Immunotherapy Strategy in Patients With Recurrent Epithelial Cancer of Ovarian, Tubal or Peritoneal Origin
Brief Title: Phase Ib/IIa Trial to Evaluate Oregovomab and Nivolumab in Epithelial Cancer of Ovarian, Tubal or Peritoneal Origin
Acronym: ORION-01
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study had poor efficacy.
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC OV-02
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Nivolumab; oregovomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab and Oregovomab (Experimental)
  Interventions: Drug: Nivolumab; Drug: Oregovomab

INTERVENTIONS:
Drug: Nivolumab — 240mg of IV Nivolumab is administered over 30 mins every 2 weeks
  Other Names: Opdivo
Drug: Oregovomab — IV Oregovomab is administered over 20 mins every 4 weeks at dose levels: 2mg, 1mg, or 0.5mg
  Other Names: OvaRex

SUMMARY:
The purpose of this study is to characterize the safety and tolerability, identify a recommended dose for expansion (RDE) / recommended phase II dose (RP2D), pharmacodynamics, and antitumor activity of Oregovomab vaccination in combination with Nivolumab as a novel combinatorial immunotherapeutic strategy in in female patients with recurrent epithelial ovarian cancer (EOC) who progressed after two or more prior lines of cytotoxic chemotherapy.

DETAILED DESCRIPTION:
This study tests the hypothesis that the combination of Oregovomab and Nivolumab will improve intracellular Cancer Antigen (CA) 125 antigen processing and elicit a stronger systemic CA 125-specific T cell response; in a manner that is synergistic, safe, and clinically efficacious in patients with relapsed EOC.

This is an open-label, single-arm, phase Ib/IIa, single-center study with dose finding and dose expansion parts.

In the phase Ib part, clinically recommended doses as monotherapy for Oregovomab (IV 2 mg Q4W, dose level 1) and Nivolumab (IV 240 mg Q2W) will be the starting doses for their combined use.

A modified "3+3" dose finding design will be employed, with 2 lower dosages of Oregovomab (dose level -1 at 1 mg Q4W; level -2 at 0.5 mg Q4W) specified in case of excessive toxicity (defined as ≥ 2 dose limiting toxicities (DLTs) out of first 3 patients, or all 6 patients) encountered at dose level 1. Three patients will be initially enrolled into dose level 1. If 0 or 1 DLT is observed, another 3 patients will be enrolled into the same dose level; otherwise de-escalate and enroll 3 patients at dose level -1. If ≤ 1 DLT is observed among the 6 patients, dose level 1 will be the RDE/RP2D of Oregovomab to be combined with Nivolumab. Likewise, in the event of de-escalation, if 0 or 1 DLT is observed at a lower dose level, a further 3 patients will be enrolled for that level; if ≤ 1 DLT is observed out of the 6 patients, that dose level will be the RDE/RP2D.

A minimum of 6 and a maximum of 18 patients will be enrolled in the dose finding part.

Approximately 14 patients are to enroll in the dose expansion part wherein they will receive Oregovomab at RDE/RP2D, combined with Nivolumab. In total, 20 patients from the dose finding and dose expansion cohorts will be treated at RDE/RP2D, and be included in the phase IIa study population.

Patients will be followed up for survival and post-progression treatment(s) over a duration of up to 36 months from the time of treatment initiation (i.e., Week 0 until up to 36 months).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   * Able to understand and voluntarily sign the Informed Consent Form (ICF). Written informed consent must be obtained before any study specific procedures that are not part of standard of care.
   * Willing and able to comply with scheduled visits, treatment schedule, laboratory test, and other protocol requirements
2. Age and Target Population

   • Age ≥ 21 years old
   * Histologically and/or cytologically confirmed diagnosis of epithelial ovarian carcinoma (serous, clear cell, endometrioid, mucinous, mixed, and others), fallopian tube and primary peritoneal carcinoma
   * Serum CA 125 level at enrollment must be at least twice the upper limit of normal (ULN) using local laboratory ranges
   * Objective evidence of disease recurrence following initial curative-intent treatment, and of progression after at least 2 prior lines of cytotoxic chemotherapy (including platinum and taxane) for advanced stage disease. Patients may have received prior treatment with Bevacizumab.
   * Presence of:

     (a) measurable disease as defined by RECIST v1.1 AND a pre-treatment serum CA 125 level ≥ 2 x ULN on 1 occasion, OR (b) non-measurable but evaluable disease such as ascites and pleural effusions attributable to disease or radiologic abnormalities that do not meet RECIST v1.1 criteria AND a pre-treatment serum CA 125 level ≥ 2 x ULN on 2 occasions at least 1 week apart, OR (c) non-evaluable, non-measurable disease as defined by RECIST v1.1 AND pre-treatment CA 125 level ≥ 2 x ULN on 2 occasions at least 1 week apart
   * Estimated life expectancy greater than 3 months
   * Performance status Eastern Cooperative Oncology Group (ECOG) 0 or 1
   * Adequate hematologic and end organ function, defined by the following local laboratory results obtained within 14 days before study entry:

     1. Absolute Neutrophil Count (ANC) ≥ 1.5 × 109/L (without granulocyte colony-stimulating factor support within 2 weeks of laboratory test used to determine eligibility)
     2. White Blood Cells (WBC) count ≥ 2.0 × 109/L
     3. Platelet count ≥ 100 × 109/L (without transfusion within 2 weeks of laboratory test used to determine eligibility)
     4. Hemoglobin ≥ 9.0 g/dL (Patients may be transfused or receive erythropoietic treatment to meet this criterion)
     5. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 30 ml/min according to Cockcroft-Gault formula below:

        Female CrCl = [(140 - age in years) x weight in kg x 1.04]/serum creatinine in mmol/L

        Male CrCl = [(140 - age in years) x weight in kg x 1.23]/ serum creatinine in mmol/L
     6. AST and ALT ≤ 3 × ULN (or ≤ 5 × ULN in patients with liver metastases)
     7. Serum bilirubin ≤ 1.5 × ULN (except patients with known Gilbert's disease who have serum bilirubin level ≤ 3 × ULN)
   * Recovery of acute AEs of prior anticancer therapies, including surgery and radiotherapy, to baseline or CTCAE grade ≤ 1 before study entry.

     * Patients with toxicities attributed to prior anticancer therapy that either are not expected to resolve and/or can result in long-lasting sequelae, such as peripheral neuropathy and ototoxicity of CTCAE grade ≤ 2 after platinum-based therapy, or are not expected to interfere with treatment on study, such as alopecia, are eligible.
3. Reproductive Status

   * Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of hCG) within 14 days before study entry.
   * No breastfeeding
   * WOCBP must agree to observe abstinence from heterosexual sexual intercourse, or use contraceptive methods that results in a failure rate of < 1% per year during the treatment period and for 5 half-lives of Nivolumab (half-life up to 25 days) plus 30 days (duration of ovulatory cycle) for a total of 23 weeks after the last IP administration. The investigator or a designated associate is requested to advise the subject on how to achieve adequate birth control.

     * A woman is considered to be of childbearing potential if she has not reached a postmenopausal state (≥ 12 consecutive months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (bilateral oophorectomy with or without hysterectomy, or bilateral tubal ligation).
     * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, properly used hormonal contraceptives that inhibit ovulation (stable on the same pill for minimum of 3 months before study entry), hormone-releasing intrauterine devices, and copper intrauterine devices.

Exclusion Criteria:

1. Cancer-specific Exclusions

   • Non-epithelial ovarian tumors, including malignant mixed Müllerian tumors (carcinosarcoma), or ovarian tumors with low malignant potential (i.e., borderline tumors).
   * Active symptomatic central nervous system (CNS) metastases. Patients with previous CNS metastases are eligible provided that they underwent CNS irradiation, are asymptomatic, do not require treatment with radiation therapy or anticonvulsants, and have stable disease at the screening tumor assessment. In addition, these patients must have been either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisolone (or equivalent).
   * Spinal cord compression not definitively treated with surgery and/or radiation. Patients with previously diagnosed and treated spinal cord compression are eligible provided that they have stable disease at the screening tumor assessment. In addition, these patients must have been either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisolone (or equivalent).
   * Leptomeningeal carcinomatosis
   * Uncontrolled pleural effusion(s), pericardial effusion, or ascites requiring recurrent drainage procedures

     o Patients with functioning pleural and/or peritoneal drainage catheters/devices in situ at time of study entry may be eligible.
   * Previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) unless a complete remission was achieved at least 2 years before study entry AND no additional therapy is required, or anticipated to be required, during the study period.
2. General Medical Exclusions

   * Pregnant or lactating women
   * Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome
   * Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months before study entry, unstable arrhythmias/heart block, or unstable angina

     o Patients with a known left ventricular ejection fraction (LVEF) < 40% or pre-existing poorly controlled hypertension (systolic blood pressure > 160 mmHg or diastolic pressure > 90 mmHg despite optimal medical management) will be excluded.
     * Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
     * Patients with stable cardiac arrhythmia requiring stable dose(s) of anti-arrhythmic therapy may be eligible.
   * Severe infections within 4 weeks before study entry including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
   * Significant traumatic injury, or major surgical procedure within 4 weeks before study entry, or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
   * History of abdominal fistula, history of gastrointestinal perforation, and signs or symptoms of bowel obstruction
   * Symptoms or radiological evidence of active bowel obstruction
   * Non-healing wound or ulcer, or bone fracture within 3 months before study entry.
   * Systemic anticancer therapy during the study, or before study entry as follows:

     (a) Cytotoxic chemotherapy: greater than the duration of the most recent cycle of the previous regimen, with a minimum of 6 weeks for nitrosoureas and mitomycin-C and a minimum of 2 weeks for all others

     (b) Biologic therapy (e.g., antibodies): up to 2 weeks

     (c) Endocrine therapy: Fulvestrant 4 weeks; Tamoxifen 2 weeks; aromatase inhibitors 2 weeks

     (d) Continuous or intermittent small molecule therapeutic: 5 times the half-life (if known), with a minimum of 2 weeks

     (e) Immunostimulatory agent (including but not limited to interferons, interleukin-2 or other cytokines): 4 weeks or 5 times the half-life (if known), whichever is shorter
     * Patients who have not recovered from therapy-related toxicities, except alopecia, peripheral neuropathy and ototoxicity (CTCAE grade ≤ 2), to baseline or CTCAE grade ≤ 1 are also excluded.
   * Extended field radiotherapy within 4 weeks, or limited field radiotherapy within 2 weeks before study entry. Patients who have not recovered from therapy-related toxicities to baseline or CTCAE grade ≤ 1 are also excluded. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease.
   * Seizure disorder requiring anti-epileptic medication
   * Renal failure requiring hemo- or peritoneal dialysis
   * Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or administration of Investigational Products (IPs), or interfere with the interpretation of safety results
   * Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
3. Exclusions Related to Investigational Products

   • Other concurrent/ongoing systemic investigational agents
   * Previous assignment to treatment during this study. Subjects permanently withdrawn from study treatment participation will not be allowed to re-enter the study.
   * History of severe allergic, anaphylactic, or other hypersensitivity reactions to murine or humanized antibodies or fusion protein
   * Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cell products or any component of the IPs
   * Prior therapy with anti-CA 125 cancer vaccine, or anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including any other antibody or immunotherapeutic drug specifically targeting T cell co-stimulation or checkpoint pathways)
   * Active, known or suspected autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Subjects with an autoimmune paraneoplastic syndrome requiring concurrent immunosuppressive treatment are excluded.

     * Patients with controlled Type 1 diabetes mellitus, autoimmune thyroid disorders who are currently euthyroid or with residual hypothyroidism only requiring hormone replacement, skin disorders (e.g., vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger may be eligible.
   * Active use of systemic corticosteroids (≥ 10mg/day prednisolone or equivalent) or other systemic immunosuppressive agents (including but not limited to prednisolone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks before study entry, or anticipated requirement for systemic immunosuppressive medications during the study.

     * Patients who have received acute, low dose, corticosteroid medications (e.g., a one-time dose of dexamethasone for nausea) may be eligible. Replacement-dose steroids in the setting of adrenocortical insufficiency (provided this is ≤ 10mg/day prednisolone or equivalent) is permitted.
     * The use of topical, inhaled, nasal and ophthalmic corticosteroids and systemic mineralocorticoids (e.g., fludrocortisone) is allowed.
   * History of solid organ allograft or allogeneic hematopoietic stem cell transplantation
   * Pre-existing Human Immunodeficiency Virus (HIV) infection, Acquired Human Immunodeficiency Syndrome (AIDS) or chronic hepatitis C infection. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients with hepatitis B (HBV) infection (defined as having a positive HBsAg test) AND undetectable HBV DNA titer are also eligible.

     o HBV DNA must be obtained in these patients before study entry. The use of antiviral therapy to attain virological response (i.e., undetectable HBV DNA titer) in HBV-infected patients is permitted.
   * Active tuberculosis
   * Administration of a live, attenuated vaccine within 4 weeks before study entry, or anticipation that such a live attenuated vaccine will be required during the study
   * Interstitial lung disease that is symptomatic or may interfere with the detection and management of suspected drug-related pulmonary toxicity.
4. Other Exclusions Criteria

   * Inability to attend or comply with treatment of follow-up scheduling

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Number of incidences and severity of Adverse Events (AE) and Serious AEs that are treatment-related, graded based on the CTCAE v4.03 | 4 weeks from the start of treatment
Overall response rate (ORR) as per Gynecological Cancer Intergroup (GCIG) criteria | Time from date of start of treatment until best overall response of CR or PR, up to 3 years
  The proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR)
Progression-free survival (PFS) as per GCIG criteria | Time from date of start of treatment to the date of the first documented progression or death due to any cause, up to 3 years

SECONDARY OUTCOMES:
ORR as per immune-related response criteria (irRC) | Time from date of start of treatment until best overall response of CR or PR, up to 3 years
  The proportion of patients with best overall response of CR or PR
Disease control rate (DCR) as per GCIG criteria and irRC | Time from date of start of treatment until best overall response of CR, PR or SD, up to 3 years
  The proportion of patients with best overall response of CR, PR or Stable Disease (SD)
ORR in EOC subtypes | Time from date of start of treatment until best overall response of CR or PR, up to 3 years
  High Grade Serous, Clear Cell, Endometrioid, Mucinous, Mixed, Others and BRCA1/2 tumors
Overall survival (OS) as per GCIG criteria | Time from date of start of treatment to date of death due to any cause, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jack Chan, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided